CLINICAL TRIAL: NCT00055029
Title: X-Linked Juvenile Retinoschisis - Clinical and Molecular Studies
Brief Title: Clinical and Genetic Studies of X-Linked Juvenile Retinoschisis
Status: Active, not recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030033; 03-EI-0033
Record Dates: First submitted 2003-02-15; First posted 2003-02-17 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Retinoschisis
Keywords: Retinoschisis; Genomic DNA; Pedigree Analysis; Genetic Analysis; Macular Degeneration; Natural History
MeSH Terms: conditions — Retinoschisis; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected males and family members: Up to 500 participants, including a minimum of 150 males diagnosed with XLRS

SUMMARY:
This study will explore the causes and eye problems of X-linked juvenile retinoschisis (XLRS), an inherited disease that causes vision loss primarily in young males. The vision loss, which worsens over time, is a result of schisis, or splitting, of the layers of the retina (tissue that lines the back of the eye). A better understanding of why and how XLRS develops might lead to improved treatments.

Patients 9 months of age and older with XLRS and females who are suspected carriers of the gene responsible for the disease (such as the mother of the patient) may be eligible for this study. Other family members of patients also may be enrolled.

Patients will undergo the following tests and procedures:

* Personal and family medical history to review past and current medical conditions and treatments, particularly regarding eye disease, and to construct a family tree.
* Eye examination to assess visual acuity (eye chart test) and examine pupils, lens, retina, and eye movements. The pupils will be dilated with drops for this examination.
* Photography of the retina to help evaluate the status of the retina.
* Specialized eye tests to evaluate color vision, field of vision, and ability to see in the dark.
* Electroretinogram (ERG) to examine what happens to the eyes after a flash of bright light. For this test, the patient sits in a dark room for 30 minutes with his or her eyes patched. Then, a small silver disk electrode is taped to the forehead, the eye patches are removed, the surface of the eye is numbed with eye drops and contact lenses are placed on the eyes. The patient looks inside a large empty bowl and then a light flashes, first in the dark and then with a light turned on inside the bowl. The contact lenses sense small electrical signals generated by the retina when the light flashes.
* Blood test to examine DNA for genetic study of XLRS.

Family members will provide a blood sample for genetic study.

DETAILED DESCRIPTION:
Objectives:

The overall goal of this protocol is to better understand the etiology of XLRS disease to facilitate further research to identify a potential treatment for the disease. The specific primary objectives of this study are to:

1. Investigate the relationship between genotype and phenotype in X-Linked Retinoschisis by correlating four phenotype severity classes with two classes of genotypes. This is the first step in developing a comprehensive genotypephenotype

   correlation.
2. Characterize the anatomical and functional characteristics of retinoschisis to refine the phenotype scale and investigate and characterize specific XLRS1 mutations to generate a well-documented genotype-phenotype correlation map.

With the opportunity to study the genotypes and phenotypes of many affected males and the genotype of family members, a secondary objective of this study will be to develop a detailed pedigree for affected families. This information may be used to develop preliminary risk estimates for potential carrier females.

Study Population:

Up to 500 participants may enroll in this study. A minimum of 150 of participants are expected to be males diagnosed with X-Linked Retinoschisis. Participants may be recruited from the NIH and also from participating off-site locations. The quality of the genetic observation is directly proportional to the number of affected individuals and genetically-different families enrolled.

Design:

This natural history, multi-center, registry study to enroll males diagnosed with X-Linked Retinoschisis and the family members of affected individuals. Onsite affected males will undergo clinical examination and have their blood drawn for genotyping. Onsite unaffected participants will undergo eye examinations. Blood may also be drawn from the onsite unaffected participants but this is not required. Sites outside of NIH are participating as referral centers to accumulate the cohort. Offsite affected male participants will forward a blood sample and records from previous eye examinations to the NEI for review and analysis. Offsite unaffected participants will forward records from previous eye examinations and may provide a blood sample although this is not required.

Outcome Measures:

The primary outcome is the categorization of the proband s genotype and phenotype and determination of the relationship between the two.

ELIGIBILITY:
* INCLUSION CRITERIA:

Eligible participants must satisfy one of the criteria below:

* Male diagnosed with X-Linked Juvenile Retinoschisis (proband). A proband will be defined as the first X-Linked Juvenile Retinoschisis diagnosed male in a given family who contacts the NIH for participation in the study; or
* Female who is a suspected carrier (i.e., mother of proband); or
* Other relative of proband including affected and unaffected males and females.

The participant (or the participant s legal guardian) understands and signs this protocol s informed consent document and minor participants between the ages of 7 and 17 must provide assent.

EXCLUSION CRITERIA:

Affected males will be ineligible for participation if:

* The participant has a significant media opacity or other obstruction precluding a complete fundus examination including retinal photography.
* The participant is unwilling or unable to contribute a blood sample for genotyping if there is not existing genetic analysis data from a documented family member.

Both affected and unaffected individuals will be ineligible for participation if:

* The participant is younger than two years (seen at the NIH) or younger than nine months (participating offsite through medical record review and blood submission).
* The participant is unable to cooperate with study procedures without anesthesia.

Ages: 9 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 500 participants may enroll in this study. A minimum of 150 of participants are expected to be males diagnosed with X-Linked Retinoschisis. Participants may be recruited from the NIH and also from participating off-site locations.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2003-05-19 (Actual)

PRIMARY OUTCOMES:
Investigate the relationship between genotype and phenotype in X-Linked Retinoschisis by correlating four phenotype severity classes with two classes of genotypes. This is the first step in developing a comprehensive genotype-phenotype correlati... | ongoing
  The overall goal of this protocol is to better understand the etiology of XLRS disease to facilitate further research to identify a potential treatment for the disease.
Characterize the anatomical and functional characteristics of retinoschisis to refine the phenotype scale and investigate and characterize specific XLRS1 mutations to generate a well-documented genotype-phenotype correlation map. | ongoing
  The overall goal of this protocol is to better understand the etiology of XLRS disease to facilitate further research to identify a potential treatment for the disease.

SECONDARY OUTCOMES:
To develop a detailed pedigree for affected families. | ongoing
  This information may be used to develop preliminary risk estimates for potential carrier females

CONTACTS AND LOCATIONS:
Overall Officials: Laryssa A Huryn, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - William Beaumont Hospital, Rochester, Michigan

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-EI-0033.html